CLINICAL TRIAL: NCT04443582
Title: An Exploratory Study of Correlating Point Of Care Ultrasound (POCUS) Measures of Sleep Apnea With STOP-BANG Scoring and Apnea-Hypopnea Index (AHI)
Brief Title: Point-of-care-Ultrasound for Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Rakesh Sondekoppam Vijayashankar (Other)
Responsible Party: Sponsor-Investigator, Rakesh Sondekoppam Vijayashankar, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202001068
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with obstructive sleep apnea (OSA) are at risk for respiratory dysfunction in the perioperative environment. The study is designed to evaluate if point-of-care-ultrasound (POCUS) measurements of upper airway anatomy may identify patients with OSA and their severity.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by recurrent collapse of the pharyngeal airway during sleep, resulting in substantially reduced (hypopnea) or complete cessation (apnea) of airflow despite ongoing breathing efforts. OSA has long been recognized as a heterogeneous disorder with potentially multiple contributing pathophysiological causes but with significant impact to perioperative morbidity. Various OSA phenotypes exist but, the predominant feature is a narrow and collapsible upper airway anatomy and is an interplay between pharyngeal soft tissue, genioglossus muscle tone and the bony anatomy and accounts for up to two-thirds of the variation in the AHI. Identification of moderate-severe OSA is crucial to prevent potential life-threatening cardiopulmonary complications perioperatively.(1) However, a large proportion of patients with OSA remain undiagnosed at the time of surgery.(2) Current screening tools are mainly questionnaire based and are largely sensitive but not specific (3) resulting in many false positives, unnecessary increased resource utilization, cost burden, and legal implications. Gold standard laboratory polysomnography(PSG) study is expensive and not widely available. Point-of-care ultrasound (POCUS) is a readily available, portable, noninvasive tool that has been used for airway evaluation and may be useful for OSA screening.(4-8) Study investigators want to evaluate the various POCUS measures of OSA in the perioperative population and correlate these measurements with the PSG based severity of OSA (based on apnea-hypopnea index -AHI) to find out the best measure or a combination of measures to diagnose the incidence and severity of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* Age 18 through 85
* History of previous sleep study polysomnography (PSG)

Exclusion Criteria:

* No prior sleep study
* History of central sleep apnea
* Craniofacial/oropharyngeal malformations
* Oropharyngeal surgery since the last sleep study
* Ear/Nose/Throat tumor
* History of Ear/Nose/Throat surgery
* Inability to consent
* Non-English speaking

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for surgeries who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of POCUS measurements with AHI and/or STOP-Bang Scores | 1 day
  The study is designed to assess if there is a correlation of one or a combination of point-of-care-ultrasound measurements with the severity of OSA as denoted by apnea-hypopnea index (AHI) from previous sleep study and/or STOP-Bang scores noted for the presence of OSA in screening exam prior to surgical procedures that require intubation.
  STOP-Bang denotes Snoring, Tired, Observed (anyone observed you stop breathing), Pressure (high blood pressure), Body mass index (more than 35 kg/m2), Age (older than 50), Neck size, Gender

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh V. Sondekoppam, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memtsoudis SG, Stundner O, Rasul R, Chiu YL, Sun X, Ramachandran SK, Kaw R, Fleischut P, Mazumdar M. The impact of sleep apnea on postoperative utilization of resources and adverse outcomes. Anesth Analg. 2014 Feb;118(2):407-418. doi: 10.1213/ANE.0000000000000051. PMID 24445639
- [Background] Singh M, Liao P, Kobah S, Wijeysundera DN, Shapiro C, Chung F. Proportion of surgical patients with undiagnosed obstructive sleep apnoea. Br J Anaesth. 2013 Apr;110(4):629-36. doi: 10.1093/bja/aes465. Epub 2012 Dec 19. PMID 23257990
- [Background] Nagappa M, Liao P, Wong J, Auckley D, Ramachandran SK, Memtsoudis S, Mokhlesi B, Chung F. Validation of the STOP-Bang Questionnaire as a Screening Tool for Obstructive Sleep Apnea among Different Populations: A Systematic Review and Meta-Analysis. PLoS One. 2015 Dec 14;10(12):e0143697. doi: 10.1371/journal.pone.0143697. eCollection 2015. PMID 26658438
- [Background] Chen JW, Chang CH, Wang SJ, Chang YT, Huang CC. Submental ultrasound measurement of dynamic tongue base thickness in patients with obstructive sleep apnea. Ultrasound Med Biol. 2014 Nov;40(11):2590-8. doi: 10.1016/j.ultrasmedbio.2014.06.019. Epub 2014 Sep 12. PMID 25220277
- [Background] Lahav Y, Rosenzweig E, Heyman Z, Doljansky J, Green A, Dagan Y. Tongue base ultrasound: a diagnostic tool for predicting obstructive sleep apnea. Ann Otol Rhinol Laryngol. 2009 Mar;118(3):179-84. doi: 10.1177/000348940911800304. PMID 19374148
- [Background] Liu KH, Chu WC, To KW, Ko FW, Tong MW, Chan JW, Hui DS. Sonographic measurement of lateral parapharyngeal wall thickness in patients with obstructive sleep apnea. Sleep. 2007 Nov;30(11):1503-8. doi: 10.1093/sleep/30.11.1503. PMID 18041482
- [Background] Shu CC, Lee P, Lin JW, Huang CT, Chang YC, Yu CJ, Wang HC. The use of sub-mental ultrasonography for identifying patients with severe obstructive sleep apnea. PLoS One. 2013 May 10;8(5):e62848. doi: 10.1371/journal.pone.0062848. Print 2013. PMID 23675433
- [Background] Siegel H, Sonies BC, Graham B, McCutchen C, Hunter K, Vega-Bermudez F, Sato S. Obstructive sleep apnea: A study by simultaneous polysomnography and ultrasonic imaging. Neurology. 2000 May 9;54(9):1872. doi: 10.1212/wnl.54.9.1872. No abstract available. PMID 10802805